CLINICAL TRIAL: NCT06281119
Title: A Phase-3b, Partially Double-blind, Randomized, Multi-country Clinical Study to Evaluate the Immunogenicity,safety, and Reactogenicity of SIIPL QHPV Vaccine (CERVAVAC®) in Women Living with HIV Aged 15-25 Years
Brief Title: Clinical Study to Evaluate SIIPL QHPV Vaccine (CERVAVAC®) in Women Living with HIV Aged 15-25 Years
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SII-qHPV/MC-03
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Human Papillomavirus Infection
Keywords: Cervavac; Quadrivalent; HPV; Vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — Clinical Protocols; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cervavac administered as three doses (Experimental): Recombinant Quadrivalent Human Papillomavirus (Types 6,11 16, 18) Vaccine manufactured by Serum Institute of India Pvt Ltd administered as three doses at day 0, 60 and 180.
  Interventions: Biological: Cervavac as three dose regimen
- Cervavac administered as two doses (Experimental): Recombinant Quadrivalent Human Papillomavirus (Types 6,11 16, 18) Vaccine manufactured by Serum Institute of India Pvt Ltd administered as two doses at day 0 and 180.
  Interventions: Biological: Cervavac as two dose regimen
- Gardasil administered as three doses (Active Comparator): Recombinant Quadrivalent Human Papillomavirus (Types 6,11 16, 18) Vaccine manufactured by MSD administered as three doses at day 0, 60 and 180.
  Interventions: Biological: Gardasil as three dose regimen

INTERVENTIONS:
Biological: Cervavac as three dose regimen — Cervavac manufactured by Serum Institute of India Pvt Ltd administered as three doses at day 0, 60 and 180.
  Arms: Cervavac administered as three doses
Biological: Cervavac as two dose regimen — Cervavac manufactured by Serum Institute of India Pvt Ltd administered as two doses at day 0 and 180.
  Arms: Cervavac administered as two doses
Biological: Gardasil as three dose regimen — Gardasil manufactured by MSD administered as a three doses at day 0,60 and 180.
  Arms: Gardasil administered as three doses

SUMMARY:
Human papillomavirus (HPV) infection is the most common viral infection of the reproductive tract. Up to 80%of the sexually active females and men will be infected with HPV at some point in their lives and some may be repeatedly infected. The main burden of HPV-related disease is due to cervical cancer. Since cervical screening only detects precancerous and cancerous changes after they have occurred, HPV vaccination is primary prevention. People with HIV infection, even when effectively treated with antiretroviral therapy (ARV),are at higher risk of acquiring infection with multiple HPV types and are also known to be predisposed to a higher risk of HPV infection and subsequent CIN lesions. Vaccination of this high-risk group with HPV vaccine is highly beneficial. SIIPL's qHPV vaccine CERVAVAC®, India's first indigenous qHPV vaccine has received marketing authorization in India. The current study is a Phase 3b study to evaluate the immunogenicity and safety of two- and three-dose schedules of SIIPL qHPV vaccine in women living with HIV (WLWH) aged 15-25years.

DETAILED DESCRIPTION:
A Phase-3b, partially double-blind, randomized, multi-country study to assess the immunogenicity, safety, and reactogenicity of SIIPL qHPV vaccine in WLWH aged 15-25 years. A total of 450 subjects will be enrolled in the study such that 150 subjects in each group receive either 3-doses of SIIPL qHPV vaccine, 2-doses of SIIPL qHPV vaccine or 3-doses of Gardasil®.

Subjects will be randomized in a 1:1:1 ratio to a 2-dose or 3-dose schedule of SIIPL qHPV vaccine or 3-dose schedule of Gardasil®. This study is designed as a partially double-blind, randomized study with a primary objective to compare the immunogenicity of the 3-dose schedule of SIIPL qHPV vaccine versus a 3-dose schedule of Gardasil®. The secondary objectives include comparison in the immune response between WLWH receiving 2-dose schedule of SIIPL qHPV vaccine and a 3-dose schedule of SIIPL qHPV. The immunogenicity data will be collected up to Month 12 and data at 7-month will be considered for analysis of primary immunogenicity endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Women Living with HIV aged 15-25 years at the time of screening
2. Subjects with age 18 years and above, should be willing and able to provide written informed consent while for subjects <18*years of age, parents willing to provide written informed consent and subject is willing to sign written assent form for participation prior to initiating any study related procedure.
3. Subject or parent willing to comply with all study requirements.
4. Subjects who are determined by medical history, physical examination and clinical judgment of the Investigator to be eligible for inclusion in the study.
5. Women of childbearing potential (WOCBP) (sexually active/ ≥18 years of age) must meet all the following criteria:

   Have practiced effective contraception (such as any one of the following: oral, transdermal, injectable or implanted contraceptive; condoms; occlusive cap [diaphragm or cervical vault caps]; spermicidal foam/gel/cream, etc.) or have abstained from all activities that could result in pregnancy from the time of screening up to first vaccine administration (Day 0).

   Have a negative Urine Pregnancy Test (UPT) at screening and on the day of vaccination (Day 0).

   Have agreed to continue effective contraception during the entire treatment period and for two months after completion of the vaccination series.
6. Subject must be asymptomatic (or only have persistent generalized lymphadenopathy) regardless of prior clinical stage.
7. If the subjects were currently taking antiretroviral (ARV) therapy, subjects were to be on highly active antiretroviral therapy (HAART), have undetectable viral load reported at least six months prior, and have a CD4+ cell count >350 cells/mm3 at study entry.
8. If the subjects are not on HAART, subjects should have a CD4+ cell count > 350 cells/mm3 at study entry.

Exclusion Criteria:

1. Known history of prior vaccination with HPV vaccine.
2. Concurrently enrolled in clinical studies of investigational agents or studies involving collection of cervical/genital specimens.
3. Current diagnosis or prior history of genital warts or treatment of genital warts.
4. Current diagnosis or history of treatment for cervical pre malignancies or malignancies.
5. Pregnant females.
6. History of any allergic diseases or severe allergic reaction to any agent.
7. Presence of an acute illness and/or fever at the time of vaccination or during the 72 hours prior to the vaccination.
8. Presence of active tuberculosis or currently on TB therapy.
9. Bleeding diathesis or uncontrolled condition associated with prolonged bleeding that would, in the opinion of the Investigator, contraindicate intramuscular injection.
10. History of major congenital defects or illness that requires medical therapy, as determined by medical history or clinical assessment.
11. History of chronic administration of high doses of corticosteroids, cytotoxic agents or radiotherapy or immunoglobulins, immunosuppressants or other immune-modifying drugs in last 3 months or planned at any time during the study.
12. History of receiving a blood transfusion or other blood products in three months prior to screening.
13. History of any major pulmonary, cardiovascular, renal, neurological, metabolic, gastro-intestinal, hepato-biliary, hematological functional abnormality, mental or physical disability, blood dyscrasia or any condition which in the opinion of the investigator might interfere with the evaluation of the study objectives.
14. History of any cancer, organ transplant or any other immune system disease (other than HIV/AIDs).
15. Subject or subject's parent, is or has an immediate family member who is study specific site staff directly involved with this trial.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Women
Enrollment: 450 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titers of anti HPV 16 and 18 IgG antibodies | at 1 month after the last dose
  GMTs of anti HPV 16 and 18 IgG antibodies in WLWH receiving 3 doses of SIIPL qHPV and 3 doses of Gardasil®

SECONDARY OUTCOMES:
Immune response (Geometric mean titers) of anti HPV 6 and 11 IgG antibodies | at 1 month after the last dose
  Geometric mean titers of anti HPV 6 and 11 IgG antibodies in WLWH receiving 3 doses of SIIPL qHPV or Gardasil
Geometric mean titers of anti HPV 6, 11, 16 and 18 IgG antibodies and Pecentage seroconversion | at 1 month after the last dose
  Geometric mean titers of anti HPV 6, 11, 16 and 18 IgG antibodies and Pecentage seroconversion in WLWH receiving 2 doses or 3 doses of SIIPL qHPV or 3 doses of Gardasil
Adverse Events | solicited AEs up to 7 days following each vaccination, unsolicited AEs from Day 0 through Month 7 and Month12 and SAEs from Day 0 through Month 7 and Month 12.
  Incidence, severity, and relationship of local and systemic solicited AEs up to 7 days following each vaccination. Incidence, severity, and relationship of unsolicited AEs from Day 0 through Month 7 and Month 12. Incidence, severity, and relationship of SAEs from Day 0 through Month 7 and Month 12.

OTHER OUTCOMES:
Geometric mean titers of anti HPV 6, 11, 16 and 18 IgG antibodies and Pecentage seroconversion | at Month 12
  Immune response to HPV types 6, 11, 16 & 18 in WLWH receiving 2 doses of SIIPL qHPV vaccine, 3 doses of SIIPL qHPV vaccine and 3 doses of Gardasil® vaccine, at Month 12.
Geometric mean titers of anti HPV 6, 11, 16 and 18 IgG antibodies and Pecentage | at Month 2 and 6
  Immune response to HPV types 6, 11, 16 & 18 after 1st dose
CD4+ cell count, HIV viral load, and HIV clinical staging | at Month 7 and Month 12
  Assessment of CD4+ cell count, HIV viral load, and HIV clinical staging in WLWH

CONTACTS AND LOCATIONS:
Overall Officials: Carla Chibwesha, Principal Investigator — Clinical HIV Research Unit, Helen Joseph Hospital, Johannesburg, South Africa; Nelly Mugo, Principal Investigator — CCR, KEMRI, Nairobi-Kenya & PHRD, Thika-Kenya; Tacilta Nhampossa, Principal Investigator — Manhiça Health Research Center - Manhiça Foundation,Manhiça
Locations (4):
- Kenya (2):
  - Centre For Clinical Research, Kemri, Nairobi
  - Partners in Health and Research Development (Phrd), Thika
- Manhiça Health Research Center - Manhiça Foundation (CISM-FM), Manhiça, Mozambique
- Clinical HIV Research Unit (CHRU), Helen Joseph Hospital, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Summary results for primary and secondary objectives
Supporting Information: Study Protocol
Time Frame: 12 Months after completion of the study
Access Criteria: Researchers who provide a methodologically sound proposal may be provided the access after Sponsor permission and if signed data-access agreements are in place.